CLINICAL TRIAL: NCT05731544
Title: A Phase 1/2 Randomized, Double-Blind, Placebo-Controlled Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, PK, and PD of BMF-219, an Oral Covalent Menin Inhibitor, in Healthy Adults and Adults With T2D
Brief Title: Study of BMF-219 in Healthy Adult Subjects and in Adult Subjects With Type 2 Diabetes Mellitus (T2D)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biomea Fusion Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COVALENT-111
Record Dates: First submitted 2022-12-26; First posted 2023-02-16 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Type 2 Diabetes Mellitus; Healthy Volunteers
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The subject and the investigator involved in the treatment or clinical evaluation of the subjects will be unaware of the group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1 SAD Cohorts (Experimental): Phase 1 SAD Cohorts with healthy adults randomized 3:1 receiving BMF-219 or placebo.
  A pair of sentinel subjects (randomly assigned 1 active drug and 1 placebo) will be dosed 48 hours prior to dosing of the remainder of subjects in each cohort.
  Interventions: Drug: BMF-219
- Phase 1 single dose food effect sub-study (Experimental): Phase 1 single dose food effect sub-study with healthy adults randomized 1:1:1:1:1:1 receiving BMF-219 or placebo fasted, with a low-fat meal, and with a high fat meal.
  Interventions: Drug: BMF-219
- Phase 1 single dose tablet PK sub-study (Experimental): Phase 1 single dose x3 PK tablet open-label sub-study with healthy adults randomized 1:1 receiving BMF-219 or placebo fasted, with a low-fat meal, and with a high-fat meal).
  Interventions: Drug: BMF-219
- Phase 2 MAD Cohorts (Experimental): Phase 2 MAD Cohorts with healthy adults (MAD 1, randomized 3:1) or adults with T2D (MAD 2-4 & 6-8, randomized 5:1) receiving BMF-219 or placebo. MAD 5 is BMF-219 only.
  Interventions: Drug: BMF-219
- Phase 2 Expansion Cohort (Experimental): Phase 2 Expansion Cohort adults with T2D randomized 3:1 ratio receiving BMF-219 or placebo.
  Interventions: Drug: BMF-219

INTERVENTIONS:
Drug: BMF-219 — Investigational Product

SUMMARY:
A Phase 1/ 2 Randomized, Double-Blind, Placebo-Controlled Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BMF-219, an Oral Covalent Menin Inhibitor, in Healthy Adult Subjects and in Adult Subjects with Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
This is a Phase 1/ 2 study that will examine the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of single and multiple dose levels of BMF-219, an orally bioavailable selective covalent inhibitor of menin, in healthy subjects and in subjects with T2D. This study will assess the effect of BMF-219 as single ascending dose (SAD) and multiple ascending dose (MAD), Expansion Cohort will explore 100mg and 200mg dose levels.

ELIGIBILITY:
Inclusion Criteria:

Healthy Subject Inclusion Criteria:

1. Males or females, age ≥18 and ≤65 years.
2. BMI ≥18 and ≤35 kg/m2.
3. Subjects are healthy on the basis of their medical history, physical examination, ECG, and routine laboratory data.
4. All subjects must be willing and able to provide written, signed informed consent and be willing and able to comply with all study procedures and tests.

Subjects with T2D: (MAD Cohorts) Inclusion Criteria:

1. Males or females, age ≥18 and ≤65 years.
2. Diagnosed with T2D within the last 15 years.
3. Treated with lifestyle management with or without at the most 3 anti-diabetic medications with a stable dose for at least 2 months prior to screening. If on metformin, the stable dose should be at least 500mg/day.
4. HbA1c ≥7.0% and ≤10.5%.
5. BMI ≥25 and ≤40 kg/m2.
6. Females are to be not pregnant, non-lactating.
7. All Subjects must be willing and able to provide written, signed informed consent and be willing and able to comply with all study procedures and tests.

Subjects with T2D: (Expansion Cohort) Inclusion Criteria:

1. Males or females, age ≥18 and ≤65 years.
2. Diagnosed with T2D within the last 7 years.
3. Treated with lifestyle management with or without at the most 3 anti-diabetic medications with a stable dose for at least 2 months prior to screening. If on metformin, the stable dose should be at least 500mg/day.
4. HbA1c ≥7.0% and ≤10.5%.
5. BMI ≥25 and ≤40 kg/m2.
6. Females are to be not pregnant, non-lactating.
7. All Subjects must be willing and able to provide written, signed informed consent and be willing and able to comply with all study procedures and tests.

Exclusion Criteria:

Healthy Subject Exclusion Criteria:

1. Evidence or history of any clinically significant disease or malignancy.
2. Mean QTcF ≥ 440 msec on triplicate ECGs. Use of medications known to significantly prolong the QT or QTcF interval.
3. History of hypertension or untreated hypertension (sitting systolic blood pressure (BP) ≥140 and diastolic BP ≥90 mm Hg).
4. Known self or family history (first-degree relative) of multiple endocrine neoplasia Type 1.
5. History of stomach or intestinal surgery or resection (except appendectomy, hernia repair, and/or cholecystectomy).
6. A history or evidence of HIV, HCV, or HBV infection at screening or active COVID-19 infection on screening.
7. Receiving an investigational intervention or having participated in another clinical trial within 30 days.
8. Currently dieting (formal weight loss program) and/or are currently using or have used within 2 months of screening any drugs for weight management.
9. Received prior menin inhibitor treatment.

Subjects with T2D (MAD Cohorts) Exclusion Criteria:

1. Type 1 Diabetes Mellitus or a secondary form of diabetes or any prior history of diabetic ketoacidosis.
2. Have had recurrence (≥2 episodes) of severe hypoglycemia (defined by the occurrence of neuroglycopenic symptoms requiring the assistance of another person for recovery) within the last 6 months prior to screening or, has a history of hypoglycemia unawareness or poor recognition of hypoglycemic symptoms as judged by the Investigator.
3. Known self or family history (first-degree relative) of multiple endocrine neoplasia Type 1.
4. Use of anti-diabetes medications (sulfonylureas, insulin, dipeptidyl peptidase-IV inhibitor [DPP-4I] [linagliptin and saxagliptin only] thiazolidinediones) within last 2 months prior to screening.
5. Fasting plasma glucose ≥255 mg/dL, fasting C-peptide <0.8 ng/mL, fasting insulin >55 μIU/mL.
6. Mean QTcF ≥450 ms. Use of medications known to significantly prolong the QT or QTc interval.
7. Fasting triglyceride ≥500 mg/dL.
8. Have an eGFR <60 mL/min/1.73 Equation at screening.
9. AST or ALT > 1.5 × ULN, bilirubin > 1.5 × ULN. Isolated GGT elevation >2.5 ULN without > 1.5 x ULN AST, ALT and/or total bilirubin but with a history of abnormal LFTs in the last 6 months or a medical history of a liver disorder should be excluded.
10. History of acute or chronic pancreatitis and serum lipase and/or amylase above 1.5 x ULN.
11. Active HBV or active HCV at screening. Known positive test, if any, prior to screening or history of HIV. An active COVID-19 infection at screening.
12. TSH >6 mIU/L or <0.4 mIU/L (on stable thyroid replacement dose for 3 months prior to screening).
13. Severe uncontrolled treated or untreated hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >90 mmHg).
14. History of stomach or intestinal surgery or resection and/or gastroparesis (except that appendectomy, hernia repair, and/or cholecystectomy will be allowed).
15. History of cirrhosis.
16. Currently dieting (formal weight loss program) and/or are currently using or have used within 2 months of screening any drugs for weight management.

Subjects with T2D (Expansion Cohort) Exclusion Criteria:

1. Type 1 Diabetes Mellitus or a secondary form of diabetes.
2. Prior history of diabetic ketoacidosis or hyperosmolar coma.
3. History of severe hypoglycemia (defined by the occurrence of neuroglycopenic symptoms requiring the assistance of another person for recovery) within the last 6 months prior to screening or, has a history of hypoglycemia unawareness.
4. Known self or family history (first-degree relative) of multiple endocrine neoplasia Type 1 (MEN1).
5. Use of any of the following anti-diabetes medications within 2 months prior to screening: sulfonylureas, insulin, and the dipeptidyl peptidase-4 inhibitors (DPP4i) linagliptin and saxagliptin (sitagliptin and other DPP4i allowed) thiazolidinones [TZD]) within last 2 months prior to screening.
6. Fasting plasma glucose ≥255 mg/dL, fasting C-peptide <0.8 ng/mL, fasting insulin >55 μIU/mL.
7. Mean QTcF interval >450 ms on triplicate ECGs. Use of prescription or over-the-counter medications known to significantly prolong the QT or QTc interval is excluded.
8. Fasting triglyceride ≥500 mg/dL.
9. eGFR<60 mL/min/1.73.
10. AST or ALT >1.5 × ULN, Total bilirubin >1.5 × ULN at screening.
11. History of acute or chronic pancreatitis and serum lipase and/or amylase above 1.5 x ULN.
12. Active HBV or active HCV at screening. Known positive test or history of HIV. An active COVID-19 infection at screening.
13. TSH >6 mIU/L or <0.4 mIU/L (on stable thyroid replacement dose for 3 months prior to screening).
14. Severe uncontrolled treated or untreated hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >90 mmHg).
15. History of stomach or intestinal surgery or resection and/or gastroparesis.
16. History of cirrhosis.
17. Currently dieting (formal weight loss program) and/or are currently using or have used within 2 months of screening any drugs for weight management.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Safety Assessments | 52 weeks
  Assessed by treatment emergent adverse events. (TEAEs), drug discontinuation due to TEAEs, serious adverse events, clinically significant laboratory, vital, and ECG evaluations.
Pharmacokinetics Assessments | 12 weeks
  Assessed by effect of fed conditions on serial and sparse pharmacokinetic data.
Change in HbA1c | 26 weeks
  Assess the change in HbA1c from baseline to week 26.

SECONDARY OUTCOMES:
To assess the effect on HbA1c | 26 Weeks
  Proportion of subjects achieving an HbA1c < 7% at Week 26.

OTHER OUTCOMES:
Exploratory: To determine the effects of BMF-219 on glycemic parameters in subjects with T2D. | Week 26
  Assess changes in plasma glucose, c-peptide, and insulin at different timepoints by both fasted and in response to OGTT.
Exploratory: To determine the impact of multiple ascending doses of BMF-219 on beta-cell function in subjects with T2D. | Week 26
  Descriptive summaries of homeostatic model assessment beta-cell function %beta and insulin resistance (HOMA-B and HOMA- IR).

CONTACTS AND LOCATIONS:
Overall Officials: Biomea Fusion Inc., Study Director — Biomea Fusion Inc.
Locations (39):
- United States (36):
  - Hope Clinical Research, Canoga Park, California
  - Ark Clinical Research, LLC, Fountain Valley, California
  - Velocity Clinical Research, La Mesa, California
  - Ark Clinical Research, Long Beach, California
  - Catalina Research Institute, LLC, Montclair, California
  - Metro Clinical Trials, San Bernardino, California
  - Southwest General Healthcare Center, Fort Myers, Florida
  - G+C Research Group, Hialeah, Florida
  - Sunbright Health Research Centers, Homestead, Florida
  - Avantis Clinical Research, Miami, Florida
  - Century Research LLC, Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - David Kavtaradze MD, Inc, Cordele, Georgia
  - Privia Medical Group, Savannah, Georgia
  - Cedar Crosse Research Center, Chicago, Illinois
  - IMA Clinical Research St. Louis, St Louis, Missouri
  - Santa Rosa Medical Centers of Nevada, Las Vegas, Nevada
  - Omera Health, Brooklyn, New York
  - IMA Clinical Research Manhattan, New York, New York
  - Carolina Research Center, Shelby, North Carolina
  - Wake Forest Health Network, LLC, Medical Plaza, Winston-Salem, North Carolina
  - Diabetes and Endocrinology Associates of Stark County, Canton, Ohio
  - Medical Care, LLC, Elizabethton, Tennessee
  - IMA Clinical Research, Austin, Texas
  - Velocity Clinical Research, Dallas, Texas
  - Zenos Clinical Research, Dallas, Texas
  - Synergy Groups Medical LLC, Houston, Texas
  - Synergy Group Medical, Houston, Texas
  - Synergy Group Medical, Missouri City, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - Diabetes & Glandular Disease Clinic, P.A., San Antonio, Texas
  - Simcare Medical Research, Sugar Land, Texas
  - Velocity Clinical Research, Waco, Texas
  - Velocity Clinical Research, Jordan, Utah
  - Manassas Clinical Research, Manassas, Virginia
- Canada (3):
  - BC Diabetes, Vancouver, British Columbia
  - Centricity Research LMC, Toronto, Ontario
  - BioPharma Services Inc., Toronto

IPD SHARING:
Plan to Share IPD: No